CLINICAL TRIAL: NCT06811090
Title: Effectiveness in Functional Recovery and Quality of Life After a Telerehabilitation Program for Patients With Ankle Fracture, Controlled Clinical Trial
Brief Title: Telerehabilitation in Patients With Ankle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Daniel Martínez Barro, MÉDICO NO FAMILIAR, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-2020-3401-024
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Ankle Fracture
Keywords: ankle fracture; tele-rehabilitation; functionality; quality of life
MeSH Terms: conditions — Ankle Fractures | interventions — Telerehabilitation; Hospitals, Rehabilitation

STUDY DESIGN:
Intervention Model Description: Tele-Rehabilitation Group (Online Exercise and Counselling) Conceptual definition: Rehabilitation service provided remotely through information and communication technologies. In this case, it will be carried out online through the Moodle platform.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital rehabilitation (Active Comparator): Rehabilitation program that will be carried out in person at the North Physical Medicine and Rehabilitation Unit. The program will be carried out by a physiotherapist and the patient will be taught: Information about the disease and self-care, Exercise module (stretching, strengthening and proprioception), gait re-education in phases.
  Interventions: Other: Hospital rehabilitation
- Tele-rehabilitation (Experimental): The Moodle application will be installed on your mobile phone to access the online content that will be integrated into three modules: 1) Information module on the disease and self-care, 2) Exercise module (stretching, strengthening and proprioception), 3) Phased walking module. Which will be integrated with video and text.
  Interventions: Other: Tele-rehabilitation

INTERVENTIONS:
Other: Tele-rehabilitation — Rehabilitation service provided remotely through information and communication technologies.
  Arms: Tele-rehabilitation
Other: Hospital rehabilitation — Rehabilitation program that will be carried out in person at the North Physical Medicine and Rehabilitation Unit. The program will be carried out by a physiotherapist and the patient will be taught: Information about the disease and self-care, Exercise module (Stretching, strengthening and proprioception), and phased gait re-education.
  Arms: Hospital rehabilitation

SUMMARY:
The objective of this clinical trial is to determine the effectiveness of a telerehabilitation program in the recovery of functionality and quality of life in patients recovering from ankle fracture. The main questions to be answered are:

What is the effectiveness of a telerehabilitation program in the recovery of functionality in patients with ankle fracture?

What is the effectiveness of a telerehabilitation program in the recovery of quality of life in patients with ankle fracture?

The researchers will compare the telerehabilitation program against the usual hospital rehabilitation procedure to see if there are differences in functional recovery and quality of life.

Participants will take a telerehabilitation program at home with the help of smartphones or will be sent to the usual hospital procedure for in-person rehabilitation.

They will have monthly in-person follow-up until 3 months, and by telephone at 6 months for the evaluation of their functionality and quality of life.

DETAILED DESCRIPTION:
Patients will be selected from the pelvic limb consultation, they will be invited to go to the tele-rehabilitation module where they will be taught the rehabilitation program that they must carry out, as well as written information about the program. Once the teaching is finished, they will be asked if they have any questions to clarify them. Once the teaching is finished, they will be followed up through the Moodle platform to see their clinical evolution and identify the date of their discharge from work. Later, this group will be compared with the patients who carried out their rehabilitation treatment in the usual way.

Randomization Randomization will be carried out through a software-based randomization program. The assignment will be done by balanced random blocks, block size 8, with an assignment ratio of 1:1. The recruitment of participants, the assignment of participants to the interventions and the evaluations will be carried out by medical evaluators.

Blinding of subjects, therapists and evaluators: Due to the nature of the intervention, it is not possible to blind participants and therapists. However, the initial and final evaluators will not be aware of the treatment group to which the study subject belongs, and the statistical analysis will be performed in a blinded manner, only the treatment will be mentioned as Group A or Group B

Data quality: Several strategies will be implemented to ensure data quality. All procedures will be adjusted with the standard operating procedures of the North Physical Medicine and Rehabilitation Unit. Evaluators and treating physiotherapists will receive appropriate training before working. Compliance with the intervention follow-up will be closely monitored by a research associate in the Physical Medicine and Rehabilitation Unit and on the platform. Forms and data processing will be periodically reviewed for accuracy. All data entry will be double-checked for accuracy.

Intervention Experimental group: Tele-Rehabilitation Group (Online Exercise and Counseling) Conceptual definition: Rehabilitation service that is provided remotely through information and communication technologies. In this case it will be carried out online through the Moodle platform.

Operational definition: The Moodle application will be installed on their mobile phone to access the online content that will be integrated into three modules: 1) Information module on the disease and self-care, 2) Exercise module (stretching, strengthening and proprioception), 3) Phased walking module. These will be integrated with video and text. Patients must log in at least 5 days a week to perform their exercises. The exercise program is based on the recommendations of national and international clinical practice guidelines, which lasts 4 weeks.

Participants will also be provided with written exercise material and a physical activity diary to assess adherence to treatment.

Control Group: Exercise supervised by the physiotherapist and advice Conceptual definition: Rehabilitation program that is carried out in person. Operational Definition: Rehabilitation program that will be carried out in person at the North Physical Medicine and Rehabilitation Unit. The program will be carried out by a physiotherapist and the patient will be taught: Information about the disease and self-care, Exercise module (stretching, strengthening and proprioception), gait re-education in phases. During the rehabilitation program, the physiotherapist can use physical means such as ultrasound, laser or interferential currents. The rehabilitation program is similar to the telerehabilitation program with a duration of 4 weeks.

Likewise, written exercise material will be provided to participants and a physical activity diary to evaluate adherence to treatment.

Statistical analysis

Descriptive statistics: qualitative variables will be summarized in absolute and relative frequencies, quantitative variables will be summarized in measures of central tendency and dispersion, if they meet the normality criterion, mean and standard deviation will be used. If they do not meet the assumption, median and interquartile ranges will be used.

Inferential statistics: For the comparison of the dependent variables between the telerehabilitation group and the traditional rehabilitation group, at the end of the study, the Student t test will be used for independent samples.

Likewise, to assess the evolution of the dependent variables in the same group, the Kruskal Wallis test will be used.

In order to identify possible confounding variables, the clinical and demographic characteristics of both groups will be compared. The Student t test will be used to compare quantitative variables and the CHi2 test will be used to compare qualitative variables. If there is a difference in any of the variables, a multivariate model will be entered to adjust the effectiveness of the intervention. A value of p< 0.05 will be considered statistically significant. All analyses will be performed on an intention-to-treat basis using the SPSS statistical program version 20.

Blind analysis Statistical analysis will be performed by a statistician who will be blinded to group assignment by dummy coding the group names. Results will be unblinded to the rest of the team once the final statistical report has been completed.

Dealing with missing data It is anticipated that missing data will be 'random'. After considering the amount and distribution of data, the likely approach will be to use multiple imputation to impute missing data for the primary outcomes. The data will be used for imputation. We did not plan to impute missing data for any of the secondary outcomes or endpoints

Sample size calculation

For the calculation of the sample size, a clinically important minimum difference of 10 points on the Ankle Functionality Scale was considered, considering a SD of 19.5, significance level of 5% and power of 80%, an estimated loss of 20% was considered, an estimated sample size of 86 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* IMSS beneficiaries treated at HTVFN for ankle fractures, over 18 years of age, discharged and referred to Rehabilitation
* WEBER A, B, and C fractures, conservative or surgical management
* Removal of immobilization
* Partial weight bearing indicated
* Access to telephone with internet (independent or with family support)

Exclusion Criteria:

Inability to complete a quality of life/functionality questionnaire Disability that limits compliance with instructions for completing a rehabilitation program at home or in an institutional setting

Elimination Criteria Loss to follow-up or individuals who wish to withdraw from the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
functionality | From admission, and with evaluations at the first, second and third month
  Rating obtained through the functional foot index. The participant rates the degree of difficulty in performing 23 different functional activities on a 10-point scale ranging from 0 ('no difficulty') to 10 ('extreme difficulty or inability to perform activity')
Quality of Life - SF-12 health questionnaire | From admission, and with evaluations at the first, second and third month
  The score obtained by the SF12 survey, which is designed to measure health-related quality of life and be the descriptive system for a multi-attribute utility instrument.
  The SF-12 response options are based on Likert-type scales that assess intensity or frequency. Each question is assigned a score, which is transformed into a scale from 0 to 100. The scores have a mean of 50 with a standard deviation of 10, so scores above or below 50 indicate better or worse health, respectively, than the reference population.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Médica de Alta Especialidad (UMAE) de Traumatología, Ortopedia y Rehabilitación "Dr. Victorio de la Fuente Narváez",, México, GUSTAVO A MADERO, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
out of respect for patient privacy

REFERENCES:
- [Background] Tenforde AS, Iaccarino MA, Borgstrom H, Hefner JE, Silver J, Ahmed M, Babu AN, Blauwet CA, Elson L, Eng C, Kotler D, Homer S, Makovitch S, McInnis KC, Vora A, Borg-Stein J. Telemedicine During COVID-19 for Outpatient Sports and Musculoskeletal Medicine Physicians. PM R. 2020 Sep;12(9):926-932. doi: 10.1002/pmrj.12422. Epub 2020 Jul 10. PMID 32424977
- [Background] Buker N, Savkin R, Ok N. Comparison of Supervised Exercise and Home Exercise After Ankle Fracture. J Foot Ankle Surg. 2019 Sep;58(5):822-827. doi: 10.1053/j.jfas.2018.11.021. PMID 31474396
- [Background] Moseley AM, Beckenkamp PR, Haas M, Herbert RD, Lin CW; EXACT Team. Rehabilitation After Immobilization for Ankle Fracture: The EXACT Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1376-85. doi: 10.1001/jama.2015.12180. PMID 26441182